CLINICAL TRIAL: NCT00003460
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Children With Primitive Neuroectodermal Tumors
Brief Title: Antineoplaston Therapy in Treating Children With Primitive Neuroectodermal Tumors
Acronym: PNET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066492; BC-BT-12 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Childhood CNS Primitive Neuroectodermal Tumor
Keywords: Recurrent primitive neuroectodermal tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Children with a primitive neuroectodermal tumor that has not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for children with primitive neuroectodermal tumors that have not responded to standard therapy provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of children with primitive neuroectodermal tumors that have not responded to standard therapy.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children (> 6 months of age) with primitive neuroectodermal tumors that has not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in children with primitive neuroectodermal tumors that has not responded to standard therapy, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in children with a brain tumor.

OVERVIEW: This is a single arm, open-label study in which children with primitive neuroectodermal tumors that have not responded to standard therapy receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (except if medically contraindicated) incurable primitive neuroectodermal tumor
* Evidence of progressive or recurrent tumor by MRI scan performed within 2 weeks prior to study entry
* Must have received and failed prior standard therapy
* Tumor must be at least 5 mm

PATIENT CHARACTERISTICS:

Age:

* 6 months to 17 years

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* No hepatic insufficiency

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No severe heart disease
* No history of congestive heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concomitant disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on a stable dose for at least 1 week prior to study entry)

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston treatment

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 1996-04; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen patients were recruited between April 1996 and January 2005. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 13
Completed | 12 (One patient was not evaluable.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: Years] | 6.1 [1.0 to 12.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 12
Participants
  Complete Response | 3
  Partial Response | 1
  Stable Disease | 1
  Progressive Disease | 7

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 13
Percentage of participants
  6 months overall survival | 61.5
  12 months overall survival | 61.5
  24 months overall survival | 53.8
  36 months overall survival | 46.2
  48 months overall survival | 38.5
  60 months overall survival | 38.5

ADVERSE EVENTS:
Time Frame: 8 years, 10 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 10/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=13)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 — The Fatigue (asthenia, lethargy, malaise) was not related to Antineoplaston therapy.
Edema/Fluid retention (General disorders) | 1 — The Edema/Fluid retention was possibly related to Antineoplaston therapy.
Infection (documented clinically): Blood (Infections and infestations) | 1 — The Infection (documented clinically): Blood was not related to Antineoplaston therapy.
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2 — The Infection (documented clinically): Lung (pneumonia) was not related to Antineoplaston therapy.
Infection with normal ANC: Lung (pneumonia) (Infections and infestations) | 1 — The Infection with normal ANC: Lung (pneumonia) was not related to Antineoplaston therapy.
Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 — The Lung (pneumonia) was not related to Antineoplaston therapy.
Middle ear (otitis media) (Ear and labyrinth disorders) | 1 — The Middle ear (otitis media) was not related to Antineoplaston therapy.
Infection: NOS (Infections and infestations) | 1 — The Infection: NOS was not related to Antineoplaston therapy.
Hypernatremia (Investigations) | 1 — The Hypernatremia was not related to Antineoplaston therapy.
Hypokalemia (Investigations) | 1 — The Hypokalemia was not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 1 — The Seizure was not related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 — One of the Somnolence/depressed level of consciousness was possibly related to Antineoplaston therapy.
Speech impairment (Nervous system disorders) | 1 — The Speech impairment was not related to Antineoplaston therapy.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 — The Dyspnea (shortness of breath) was not related to Antineoplaston therapy.
Thrombosis/thrombus/embolism (Vascular disorders) | 1 — The Thrombosis/thrombus/embolism was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=13)
Allergic reaction/hypersensitivity (including drug fever) (General disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Supraventricular and nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 1
Central venous catheter infection (Infections and infestations) | 2
Non-functional central venous catheter (General disorders) | 2
Central venous catheter: Other (General disorders) | 2
Central venous catheter: Thrombosis/embolism (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8
Fever (General disorders) | 2
Rigors/chills (General disorders) | 4
Weight gain (General disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 5
Cushingoid appearance (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 7
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 2
Infection (documented clinically): Blood (Infections and infestations) | 3
Infection (documented clinically): Bronchus (Infections and infestations) | 1
Infection (documented clinically): Eye NOS (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 3
Infection (documented clinically): Middle ear (otitis) (Infections and infestations) | 4
Infection (documented clinically): Mucosa (Infections and infestations) | 5
Infection (documented clinically): Stomach (Infections and infestations) | 2
Infection (documented clinically): Upper airway (Infections and infestations) | 3
Infection with normal ANC: Lung (pneumonia) (Infections and infestations) | 1
Infection: NOS (Infections and infestations) | 1
Infection: Skin (Infections and infestations) | 1
Hypertrychosis (Skin and subcutaneous tissue disorders) | 1
Alkaline phosphatase (Investigations) | 2
Hyperglycemia (Infections and infestations) | 2
Hypernatremia (Investigations) | 4
Hypocalcemia (Investigations) | 2
Hypoglycemia (Investigations) | 3
Hypokalemia (Investigations) | 12
Hypomagnesemia (Investigations) | 3
Hyponatremia (Investigations) | 1
Hypophosphatemia (Investigations) | 2
SGOT (Investigations) | 3
SGPT (Investigations) | 2
Uric acid, serum-high (hyperuricemia) (Investigations) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 5
Somnolence/depressed level of consciousness (Nervous system disorders) | 7
Speech impairment (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Diplopia (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain: Head/headache (Nervous system disorders) | 6
Pain: Joint (Musculoskeletal and connective tissue disorders) | 2
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Incontinence, urinary (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No